CLINICAL TRIAL: NCT04082598
Title: Antibiotic Therapy in Erupted Tooth Extractions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Antonio Barone (Other)
Responsible Party: Sponsor-Investigator, Antonio Barone, Associate Professor ( DDS, PhD, MSc), University of Pisa
Organization: University of Pisa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AB0001
Record Dates: First submitted 2019-08-14; First posted 2019-09-09 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Tooth Extraction; Post-Op Complication; Amoxicillin
Keywords: tooth extraction; antibiotics; probiotics; tooth infection; complications
MeSH Terms: conditions — Postoperative Complications | interventions — Amoxicillin-Potassium Clavulanate Combination; Lactoferrin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tooth extraction and antibiotic treatment (Experimental): Tooth extraction and Amoxicillin- clavulanic acid 875/125 mg, twice a day, for 6 days
  Interventions: Drug: Amoxicillin Clavulanate
- tooth extraction and antibiotic treatment + dietary supplement (Experimental): Tooth extraction and Amoxicillin- clavulanic acid 875/125 mg, twice a day, for 6 days + Bifidobacterium longum and Lactoferrin twice a day for 6days
  Interventions: Drug: Amoxicillin Clavulanate; Dietary Supplement: Bifidobacterium longum and Lactoferrin
- Tooth extraction (No Intervention): tooth extraction without antibiotics and/or Bifidobacterium longum and Lactoferrin

INTERVENTIONS:
Drug: Amoxicillin Clavulanate — tooth extractions are performed for all groups and antibiotics prescribed according to the allocation to the different arms
  Arms: Tooth extraction and antibiotic treatment; tooth extraction and antibiotic treatment + dietary supplement
Dietary Supplement: Bifidobacterium longum and Lactoferrin
  Arms: tooth extraction and antibiotic treatment + dietary supplement

SUMMARY:
Evaluation of the efficacy of amox+clav and of a probiotic after tooth extraction. the aim is to evaluate efficacy of antibiotic therapy after tooth extractions in preventing infections as compared to no therapy, and efficacy of probiotics in preventing gastro-intestinal adverse effects during the antibiotic treatment. The number of patients to be included is 150. The study products are: Amoxicillin + Clavulanic Acid and Bifidobacterium Longum and Lactoferrin.

DETAILED DESCRIPTION:
The main objective of this trial is to evaluate the efficacy of the antibiotic after tooth extraction in preventing infections and to evaluate the effect of probiotic in reducing the possible antibiotic side effects. In order to analyze the effect of the antibiotic in terms of patient's general discomfort, a tailored form was prepared (Appendix A). The local signs and symptoms to evaluate are swelling, pain (assessed by the Visual Analogic Scale), presence of abscess, fever, post-extraction dental alveolitis (dry socket) and presence of trismus assessed as maximal mouth opening variation (mm). In addition adverse post-extraction events will be evaluated as follows: chewing impairments (assessed by the Visual Analogic Scale), speaking impairments (assessed by the Visual Analogic Scale), daily oral hygiene maneuvers impairments (assessed by the Visual Analogic Scale) and daily activities alterations (days-off from job/study). Moreover, the patients will be provided with a painkiller's prescription and they are required to take note of the painkillers needed during the first 7 days, i.e. until the first time point recall. The prescribed painkillers will be Ibuprofen 600 mg or naproxen sodium 500mg for those patients who reported allergy to ibuprofen. Finally, it will be a researcher duty to ask the patients if they needed to assume painkillers beyond the 7th day. Since the post-surgical sequelae depend also on the difficulty of extraction, the Appendix A provides a table in which the surgeon can take note of the type of extraction.

ELIGIBILITY:
Inclusion Criteria:

* Patients who needed tooth extractions
* Patients older than 18 years
* Patients able to understand and to sign a consent form

Exclusion Criteria:

* General contraindications to oral surgery
* Third molar or impacted tooth extractions
* Patients treated or under treatment with immunosuppressive agents or patients immunocompromised
* Patients treated or under therapy with amino-bisphosphonate and anti-angiogenetic intravenous medications
* Patients who received head and neck irradiation treatments
* Patients who were diagnosed with uncontrolled diabetes
* Patients suffering from renal failure
* Pregnancy and breastfeeding patients
* Patients diagnosed with drug and alcohol addiction
* Patients who suffer from psychiatric disorders
* Patients diagnosed with allergy to penicillin and probiotic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Rate of post-operative infection after tooth extractions | 21 days
  infection, presence or absence of pus drainage
Rate of post-operative alveolar osteitis after tooth extractions | 21 days
  alveolar osteitis, presence or absence of exposed bone

SECONDARY OUTCOMES:
gastrointestinal symptoms | 21 days
  presence of abdominal pain, abdominal distension, nausea, vomit, acid reflux, gastric acidity, gastric pain, intestinal pain, gastric distension, intestinal distension and diarrhea

IPD SHARING:
Plan to Share IPD: No